CLINICAL TRIAL: NCT06315855
Title: F.L.O.S.S. Project (Facilitated Lessons on Oral and Systemic Health in Survivors)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00007140
Record Dates: First submitted 2024-02-15; First posted 2024-03-18 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Oral Mucositis; Periodontal Diseases; Cancer
MeSH Terms: conditions — Stomatitis; Periodontal Diseases; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth Intervention (THI) arm (Experimental): The THI is a 6-month intervention. Participants randomized to THI arm will engage in 6,1-hour virtual sessions with trained study personnel. Modules contain a 1) participant check-in, 2) content designed to build oral health literacy and self-efficacy, 3) and goal-setting.
  Coaches will use a facilitation guide, layered with motivational interviewing to conduct telehealth sessions. Participants will also receive biweekly text messages aligned with module content. Post-intervention follow-up will occur at 6- and 12-month post-randomization.
  Interventions: Behavioral: Telehealth Intervention (THI)
- Usual Care (UC) arm (No Intervention): This group will receive biweekly text messages on general health behaviors as a retention strategy. This arm will receive no other outside interventions. The Dental Resource directory will be provided to all participants.

INTERVENTIONS:
Behavioral: Telehealth Intervention (THI) — The THI is a 6-month intervention. On a monthly basis, the survivor will be queried via telehealth (zoom or smart phone) oral and health related symptoms by nurse practitioner or navigator. Based on the initial imaging and the monthly assessments, the patients will be provided with tools and instructions for oral health maintenance which may consist of mucositis management and/or diet and lifestyle counseling. All participants will be provided a Resource directory that is to be used to identify a dentist that is best suited for him/her. Post intervention, follow-up assessments will be conducted at 6-, 9- and 12-months post randomization.
  Arms: Telehealth Intervention (THI) arm

SUMMARY:
The investigators will conduct a 2-arm 6-month randomized clinical controlled trial to evaluate the effectiveness of an oral Telehealth Intervention (THI) in preventing cancer-related oral complications, improving oral health maintenance and oral health related quality of life, and reducing systemic inflammation compared to Usual Care (UC) among unselected cancer survivors.

DETAILED DESCRIPTION:
The goal of this study is to assess the efficacy of a Telehealth Intervention (THI) in 1) yielding more favorable oral health outcomes (e.g., reduced treatment-related mucositis, reduced gingival inflammation, tooth preservation); better oral health-related quality of life (OHRQoL). The investigators will also assess the efficacy of THI in yielding decreased systemic inflammation compared to usual care (UC).

The Study population will comprise 100 unselected cancer survivors who will be recruited through community-based approaches. The goal is to enroll 50 active treatment and 50 post-treatment into the study.

Intraoral Imaging All participants, prior to randomization will undergo an intraoral imaging assessment.

Intraoral imaging will be conducted on all study participants at the time of their baseline in- person visit. Photos of the mouth, teeth, and gums will be captured and saved in individual patient files for research and data purposes only. The images captured by the intraoral imaging exam will not be uploaded to any electronic healthcare records for dentist or hygienist use; these images are strictly for the use of research staff. These images will be the data for the study, as both baseline and succeeding follow-up images will be taken. These images will be used to analyze the oral health and overall quality of life of the subjects. The investigators will have a dental consultant review images and provide summary data.

Biospecimens Saliva samples will be collected at baseline, 6-,and 12-month post-randomization.

Participants will self-collect the saliva sample using the Omnigene Saliva DNA and RNA device (OMR-610). Blood samples (10 mL) for biomarker assessments at baseline and follow-up visits (i.e., 6- and 12- months) Inflammation markers including C-reactive protein, IL-1, IL-6, and TNF-alpha will be measured. Samples will be processed within two hours and stored at -70°C. Saliva samples will be stored for up to 21 days at room temperature, and then will be stored at -20 °C. Human and microbial DNA and RNA will be extracted to examine oral microbiome.

Survey Instruments Basic demographics and lifestyle characteristics will include smoking, physical activity, and diet, clinical characteristics, cancer-treatment questionnaire, EORTC oral and overall quality of life questionnaires (QLQ-C30 and OH-15), Oral Health Impact Profile (OHIP-14), patient-reported oral mucositis symptom scale, and Area Deprivation Index.

Anthropometric measures of height, weight, waist and hip circumference will also be collected. All survey and anthropometric measurements will be collected at baseline, 6- and 12- month post-randomization.

Clinical Trial Arms This is a six-month 2-arm randomized controlled trial comprising a Telehealth Intervention (THI) arm and a Usual Care (UC) arm as described below

Telehealth Intervention (THI) This is based on e-Health and mobile Health and utilizes the use of information and communication technologies for health. More specifically this telehealth method is a medical and public health practice that is supported by mobile devices, such as mobile phones, patient monitoring devices, personal digital assistants, and other wireless devices. This method allows for the monitoring of oral health conditions and alert the patient or oncologist about an emerging oral health issue. Moreover, telehealth reduces the need to come into an office for a visit.

Outcomes

The following outcomes will be measured in all participants at baseline and repeated at 6 and 12 months:

ORAL HEALTH OUTCOMES

1. mucositis: clinical via intro-oral imaging using the WHO oral mucositis grading scale) and the patient-reported oral mucositis symptom scale (PROMS) questionnaire
2. gingival inflammation and periodontal disease: Modified Gingival Index based on intraoral imaging
3. tooth decay: Delayed, Missing, Filled Teeth (DMFT) index based on intraoral imaging
4. oral health related quality of life: Oral health Impact Profile (14-item OHIP-14 questionnaire) and the cancer specific oral health questionnaires (EORTC Quality of Life Questionnaires - oral health)

SYSTEMIC OUTCOMES

1. systemic inflammation: Inflammation markers measured in peripheral blood samples
2. overall health related quality of life: measured using EORTS QLQ-C30 questionnaire
3. comorbidities: cardiovascular and metabolic comorbidities including diabetes, hypertension, heart disease, and stroke will be determined from the medical record

Statistical Analysis Demographic and other baseline data including cancer-related clinical characteristics will be listed and summarized descriptively by intervention arm (THI and UC). Categorical data will be presented as frequencies and percentages. For continuous data, mean, standard deviation, median, minimum, and maximum will be presented. For selected parameters, 25th and 75th percentiles will also be presented.

Intention to treat (ITT) analysis will be performed for all participants who enrolled and randomly allocated to one of the clinical trials arms to which they were randomized. Descriptive statistics will be used to summarize the original scores for the outcomes (oral and systemic health outcomes), as well as change from baseline, at each scheduled assessment timepoint for the THI and UC group. Additionally, change from baseline in the scale and subscale values at the time of each assessment will be summarized. Participants with an evaluable baseline score and at least one evaluable post baseline score during the treatment period will be included in the change from baseline analyses.

The number of participants completing each questionnaire and the number of missing or incomplete assessments will be summarized by treatment group for each scheduled assessment timepoint. A repeated measurement analysis model for longitudinal data will be used to estimate differences in the scores of mucositis, oral and systemic inflammation, tooth decay, and oral and overall quality of life between the THI and UC arms. The differences in least square means between the treatment arms and corresponding 95% confidence interval at selected timepoints will be presented. Details, including handling of missing data, will be specified in the detailed protocol for the study.

ELIGIBILITY:
Inclusion Criteria:

* male and female cancer survivors who are either ≥ 6 months after competing primary therapy for cancer treatment (N=100)
* between 25-75 years of age
* all race/ethnic groups
* own a smart phone.

Exclusion Criteria:

* all head and neck/oral cancer survivors
* less then 25 years and older than 75 years of age
* recurrence/second cancers or undergoing treatment
* unable to provide informed consent.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2026-08-25 (Estimated); Study Completion 2027-08-25 (Estimated)

PRIMARY OUTCOMES:
mucositis | baseline and repeated at 6 and 12 months
  The World Health Organization Oral Toxicity Scale rates the anatomical, and function aspects of oral mucositis. The severity of oral ulcers and ability to consume food and liquid is reported on a scale of 0 (no presentation of symptoms) to 4 (not able to tolerate food or liquid diet). Higher scores indicate worse oral mucositis symptomology.
  The PROMS questionnaire: Respondents will indicate their level of oral mucositis symptoms on a sliding scale ranging from no experience of a mucositis-related symptoms to complete experience of symptoms. Higher scores indicate worse self-reported mucositis.
gingival inflammation and periodontal disease | baseline and repeated at 6 and 12 months
  Using the modified gingival index, the investigators will rate inflammation of gums on a 5-point Likert Scale ranging from 0 (absence of inflammation) to 4(severe inflammation, marked redness, edema. Higher scores indicate more severe inflammation.
tooth decay | baseline and repeated at 6 and 12 months
  Delayed, Missing, Filled Teeth (DMFT) index based on intraoral imaging The DMFT index will be calculated by summing the number of delayed, missing, or filled teeth and dividing this value by the sum of the DMFT values in the study sample. Higher values equate to poorer tooth retention.
oral health related quality of life | baseline and repeated at 6 and 12 months
  Oral health Impact Profile (14-item OHIP-14 questionnaire) and the cancer specific oral health questionnaires (EORTC Quality of Life Questionnaires - oral health)
  This measure assesses the impact of oral health on overall wellbeing. Respondents will indicate their agreement with a statement (Yes/No). Higher scores indicate a greater impact of oral health on daily life.
  EORTC- Quality of Life Questionnaires Oral health: For items 1-11, Respondents indicate agreements on a 4-point Likert scale ranging from 1(not at all) to 4(Very much). On items 12-15, respondents indicate dichotomous agreement (Yes/No). Scores are summed and logged transformed to 0-100 scale. Higher scores indicate a better oral health related quality of life and better functioning.

SECONDARY OUTCOMES:
systemic inflammation | baseline and repeated at 6 and 12 months
  Blood samples will be processed to separate plasma and buffy coat aliquots within two hours and stores at -80 degrees Celsius. The following biomarkers will be identified: C-reactive protein (mg/dL), IL-1 (pg/mL), IL-6 (pg/mL), and TNF-alpha (pg/mL).
overall health related quality of life | baseline and repeated at 6 and 12 months
  EORTC Quality of Life-C30 will assess health-related quality of life. For items 1-28, respondents will indicate agreement on a 4-point Likert scale ranging from 1(Not at all) to 4(very Much). For items 29 and 30, respondents rate agreement on a 7-point Likert scale ranging from 1(very poor) to 7(excellent). Scores are summed and logged transformed to 0-100 scale. Higher scores indicate a better health-related quality of life and better functioning.
comorbidities | baseline and repeated at 6 and 12 months
  Captured via self-report survey, participants will indicate prior or current diagnoses of cardiovascular and metabolic comorbidities including diabetes, hypertension, cardiovascular disease, stroke, etc.
  - Anthropometrics
  * Height in centimeters rounded to the nearest tenth.
  * Weight in kilograms, captured on a calibrated scale.
  * Waist circumference in centimeters
  * Hip circumference in centimeters.

CONTACTS AND LOCATIONS:
Locations (1):
- Georgetown Lombardi Office of Minority Health, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dash C, Smith DI, Williams N, Leby C, Nyirenda N, Makambi KH, Adams-Campbell L. The FLOSS Project: study protocol for a parallel-group, two-arm randomized controlled trial examining the efficacy of telehealth in promoting oral and systemic health in cancer survivors. Trials. 2025 Nov 24;26(1):535. doi: 10.1186/s13063-025-09247-1. PMID 41286997